CLINICAL TRIAL: NCT02993055
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ulimorelin (LP101)
Brief Title: A Study to Assess Ulimorelin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lyric Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP101-CL-101
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ulimorelin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ulimorelin (Experimental): Active
  Interventions: Drug: Ulimorelin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ulimorelin
  Arms: Ulimorelin
Other: Placebo
  Arms: Placebo

SUMMARY:
A Phase I dose escalation study involving healthy subjects.

ELIGIBILITY:
Inclusion Criteria

1. Ethics committee approved written informed consent and privacy language per national regulations must be obtained from the subject before any study-related procedures (including withdrawal of prohibited medication, if applicable)
2. Subject is a healthy male or non-pregnant (as documented by a negative urine pregnancy test at screening and admission to the clinical study unit on Day -1 of the SAD phase and Day -3 of MAD phase), non-lactating healthy female who is aged between 18 and 55 years, inclusive, weighs between 50 kg to 90 kg, and has a body mass index in the range of 18 to 35 kg/m2 or, if outside the range, considered not clinically significant by the investigator
3. Subject is a non-smoker and has not used tobacco for a minimum of 6 months before screening (a breath carbon monoxide reading of ≤10 ppm at screening)
4. Subject must be willing and able to communicate and participate in the whole study
5. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subject has clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator at screening or admission as determined by the investigator
2. Subject has abnormal and clinically significant 12-lead ECG at screening or on admission to the clinical study unit at each period
3. Subject has 12-lead ECG demonstrating QTcF >450 msec in males and >470 msec in females at screening. If QTcF exceeds these limits, the ECG should be repeated 2 more times at least 1 minute apart, and the average of the 3 QTcF values should be used to determine the subject's eligibility
4. Subject has a known serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
5. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
6. Subject has supine blood pressure or pulse rate outside of the ranges 90 to 140 mmHg systolic blood pressure/40 to 90 mmHg diastolic blood pressure and 50 to 90 bpm, respectively, at screening or admission or a heart rate below 46 bpm at pre-dose on Day 1 of either the SAD or MAD phase
7. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
8. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 2 g per day paracetamol) or herbal remedies in the 7 days before IMP administration
9. Subject has received a vaccine within 30 days before first dosing
10. Subject has a history of drug or alcohol abuse within the past 2 years before screening or a positive result for alcohol at screening or admission
11. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 1⁄2 pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
12. Positive drugs of abuse test result
13. Subject has a history of any clinically significant neurological, GI (especially prior gastric or oesophageal surgery, gastroparesis, peptic ulceration, GI bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome), renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine (diabetes mellitus), respiratory or haematological disorder or disease or any other medical condition that, in the opinion of the investigator, would preclude participation in the study
14. Subject has participated in another investigational study within the past 3 months before study drug administration, or subject has previously participated in a study with ulimorelin
15. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
16. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
17. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
18. Donation or loss of greater than 400 mL of blood within the previous 3 months
19. History of upper GI surgery
20. Acute diarrhoea or constipation in the 7 days before the predicted first study day. If screening occurs >7 days before the first study day, this criterion will be determined on first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
21. Subject has any other condition that in the opinion of the investigator precludes participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Measuring the Cmax after administration of Ulimorelin | 7 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] James J, Mair S, Doll W, Sandefer E, Wurtman D, Maurer A, Deane AM, Harris MS. The effects of ulimorelin, a ghrelin agonist, on liquid gastric emptying and colonic transit in humans. Neurogastroenterol Motil. 2020 Mar;32(3):e13784. doi: 10.1111/nmo.13784. Epub 2020 Feb 3. PMID 32017341